CLINICAL TRIAL: NCT05035953
Title: Effect of Thrombolysis Combined With Edaravone Dexborneol for Acute Ischemic Stroke Patients: a Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Thrombolysis Combined With Edaravone Dexborneol on Hemorrhagic Transformation for Acute Ischemic Stroke
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Huashan Hospital (Other)
Collaborators: Shanghai Stroke Association (Unknown)
Responsible Party: Principal Investigator, Qiang Dong, MD, PhD, Director of Neurology Department, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SMA-AIS-003
Record Dates: First submitted 2021-09-03; First posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Stroke, Ischemic
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Edaravone (Experimental): Edaravone Dexborneol injection
  Interventions: Drug: Edaravone Dexborneol
- Placebo (Placebo Comparator): Edaravone Dexborneol matching injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Edaravone Dexborneol — Edaravone Dexborneol 37.5 mg (containing Edaravone 30 mg and Dexborneol 7.5 mg), BID, 14 days, addition to thrombolysis
  Arms: Edaravone
Drug: Placebo — Edaravone Dexborneol matching injection, addition to thrombolysis
  Arms: Placebo

SUMMARY:
To explore the safety and efficacy of edaravone dexborneol for the treatment of acute ischemic stroke patients who received thrombolysis.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke;
* 18 to 80 years of age;
* There are clear signs of neurological deficit: 8≤NIHSS score≤24;
* Received alteplase thrombolysis therapy within 4.5 hours after onset;
* Patients signed written inform consent

Exclusion Criteria:

* Patients need endovascular therapy or bridge therapy;
* Cranial CT scan finds intracranial bleeding disorders: hemorrhagic stroke, epidural hematoma, intracranial hematoma, intraventricular hemorrhage, subarachnoid hemorrhage;
* Severe head trauma or stroke, intracranial tumor or large intracranial aneurysm within 3 months;
* Intracranial or intraspinal surgery within 3 months;
* Active visceral hemorrhage
* Major surgery within 2 weeks or arterial puncture within 1 week that is difficult to compress the hemostatic site;
* Unknown onset time;
* Rapid improvement of symptoms or mild symptoms before thrombolysis therapy;
* A platelet count below 100,000/mm3 indicates a propensity for acute bleeding;
* Therapeutic neuroprotective agents have been applied after onset of stroke, including commercially available edaravone, nimodipine, ganglioside, citicoline, piracetam, butyl benzene peptides, Urinary Kallidinogenase;
* Patients with severe mental disorders and dementia;
* ALT or AST is greater than 2.0×ULN or previously known liver diseases, such as acute hepatitis, chronic active hepatitis, liver cirrhosis;
* Serum Creatinine (SCr) is greater than 1.5×ULN, Creatinine Clearance (CrCl) is less than 50 ml/min or previously known severe renal diseases;
* Patients with malignant tumors or severe systemic disease;
* allergic to edaravone , (+)-Borneol or related excipients;
* Pregnant or lactating women;
* Have major surgery within 4 weeks before enrollment;
* Participated in other clinical studies within 30 days before randomization; or participating in other clinical trials at present;
* The investigators consider the patients are not suitable for this trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-09-13 (Estimated); Primary Completion 2023-09-13 (Estimated); Study Completion 2024-03-13 (Estimated)

PRIMARY OUTCOMES:
The proportion of symptomatic intracranial hemorrhage | 36-48 hours

SECONDARY OUTCOMES:
The proportion of symptomatic intracranial hemorrhage | 7 days
The proportion of intracranial hemorrhage | 36-48 hours, 7 days
The proportion of Participants With modified Rankin Scale (mRS) Score 0 to 1 | 90 days
The change in the NIH stroke scale (NIHSS) from the baseline | 36-48 hours, 7, 14 and 90 days
The proportion of Participants With Barthel Index (BI) score greater than or equal to 95 | 14 and 90 days
Vascular recanalization | 36-48 hours
Blood Brain Barrier Permeability | 36-48 hours
Proportion of Encephaledema | 36-48 hours
Proportion of Death | 90 days

IPD SHARING:
Plan to Share IPD: Undecided